CLINICAL TRIAL: NCT03415828
Title: Intradiscal Gelified Ethanol Versus Intradiscal Steroid in Refractory Lumbar Discogenic Pain: a Randomized Single-blind Study
Brief Title: Ethanol Gel Versus Steroid in Refractory Lumbar Discogenic Pain
Acronym: IDIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gelscom SAS (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-A03259-44
Record Dates: First submitted 2018-01-09; First posted 2018-01-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Discogenic Pain (Disorder)
MeSH Terms: interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethanol gel (Experimental): CE-marked medical device used according to its instructions for use: GELSCOM® Single injection in the selected disc(s) of 0.6 to 2.2 ml
  Interventions: Device: Ethanol gel
- Steroid infiltration (Active Comparator): Authorized drug used according to its summary product characteristics: HYDROCORTANCYL 2,5 POUR CENT Single injection in the selected disc(s) of 0.2 to 2.0 ml
  Interventions: Drug: Prednisolone acetate

INTERVENTIONS:
Device: Ethanol gel — Intradiscal injection of ethanol gel
  Other Names: DISCOGEL®
  Arms: Ethanol gel
Drug: Prednisolone acetate — Intradiscal infiltration of steroids
  Other Names: HYDROCORTANCYL 2,5 POUR CENT
  Arms: Steroid infiltration

SUMMARY:
DISCOGEL® is on the market since 2007. About 20,000 kits were sold to date (October 2017). The device re-obtained its CE mark in 2017.

A clinical evaluation was performed by bibliographic route in 2016. Clinical data on more than 600 patients treated by DISCOGEL® were analyzed. These data should be confirmed by monitoring on the long term, with a large cohort of patients, over a two-year follow-up period.

As part of the post-CE surveillance, the manufacturer GELSCOM is responsible of this "Post-Market Clinical Follow-up" (PMCF) study in accordance with Directive 93/42/EEC and MEDDEV guide 2.12/2, to assess the efficacy and the long-term safety of DISCOGEL®.

The study is comparative. The results will evaluate the performance and safety of the CE-marked medical device used in "real life", in comparison with a steroid infiltration, used according to its indication and to the current standards. It will include economic data. Patients and evaluators will be blinded. Both DISCOGEL® and HYDROCORTANCYL 2,5 POUR CENT are authorized products used according to their intended use.

This is an interventional, prospective, national, multi-center, comparative, randomized, single-blind (patient and evaluator) post-market clinical study. The primary objective is to compare the short-term efficacy profile of DISCOGEL® versus intradiscal steroid.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older;
* 2-month refractory pain to conservative treatment, non-surgical patients;
* Chronic discogenic pain (1 or 2 lumbar discs) with concordant MR imaging;
* Symptomatic for at least 8 weeks despite appropriate medical treatment;
* Patient who agrees to participate in the study and who signed the informed consent form;
* Patient with social protection.

Exclusion Criteria:

* Previous surgical treatment of the studied disc(s);
* Patient with pure radicular pain;
* Sick leave of more than 12 months secondary to the symptoms;
* Patients who cannot read or write French;
* History of cognitive-behavioral disorders that could interact with assessment by self-questionnaire;
* Local or general infection, or suspicion of infection;
* Severe coagulation disorders;
* Other rheumatic inflammatory disease;
* Undercurrent serious pathology with life expectancy < 2 years;
* Female of childbearing age that are known to be pregnant during inclusion visit or wishing to become pregnant before treatment;
* Subject who has forfeited their freedom by administrative or legal award, or is under guardianship or under limited judicial protection
* Patient participating in another interventional clinical trial or testing an experimental drug within 30 days of inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
Short-term efficacy profile | Month 3
  Compare the short-term efficacy profile of DISCOGEL® versus intradiscal steroid: percentage of patients with a pain relief defined by a Low Back Pain (LBP) intensity<4 cm on a Local Verbal Rating Scale (0 = no pain to 10 = maximum imaginable pain)

SECONDARY OUTCOMES:
Long-term efficacy profile | Month 12
  Compare the long-term efficacy profile of DISCOGEL® versus intradiscal steroid: Local Verbal Rating Scale: on back, bottom, thigh, leg, foot
Long-term efficacy profile | Month 24
  Compare the long-term efficacy profile of DISCOGEL® versus intradiscal steroid: Local Verbal Rating Scale: on back, bottom, thigh, leg, foot
Short-term safety profile | Month 3
  Analyze the short- and long-term safety profile of DISCOGEL®: rates of complications and adverse reactions
Long-term safety profile | Month 12
  Analyze the short- and long-term safety profile of DISCOGEL®: rates of complications and adverse reactions
Long-term safety profile | Month 24
  Analyze the short- and long-term safety profile of DISCOGEL®: rates of complications and adverse reactions
Questionnaire OSWESTRY | Month 24
  Describe the rate of subjects improved 24 months after treatment: OSWESTRY scale
Questionnaire MacNab | Month 24
  Subjective improvement 24 months after treatment: MacNab scale
Radiography | Month 3
  Describe radiologic evolution of the lesions: radiography of the herniated disc
Radiography | Month 12
  Describe radiologic evolution of the lesions: radiography of the herniated disc
Radiography | Month 24
  Describe radiologic evolution of the lesions: radiography of the herniated disc
Magnetic Resonance Imaging | Month 3
  Describe radiologic evolution of the lesions: MRI of the herniated disc
Procedures costs | Day 0
  Compare the cost linked to the DISCOGEL® procedure and the cost linked to a steroid infiltration or surgery
Procedures durations | Day 0
  Compare the duration of the treatment procedures between a DISCOGEL® injection and a steroid infiltration or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu de Sèze, Dr, Study Chair — CHU Bordeaux Pellegrin
Locations (5):
- France (5):
  - Hospital Pellegrin, Bordeaux
  - Hospital St-Dié-des-Vosges, Saint-Dié
  - Hospital SUD La Reunion, Saint-Pierre
  - Hospital St-Etienne, Saint-Priest-en-Jarez
  - Hospital Valence, Valence

IPD SHARING:
Plan to Share IPD: No